CLINICAL TRIAL: NCT04190589
Title: A Single Center Prospective Study Comparing Robot-assisted and Open Operation With Complete Mesocolic Excision (CME) in Extended Right Colectomy for Colon Cancer in the Right Flexure and Transverse Colon
Brief Title: Prospective Study of Extended Robotic Right Hemicolectomy With Complete Mesocolic Excision for Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RobotCME01
Record Dates: First submitted 2019-12-02; First posted 2019-12-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Robot; Hemicolectomy; Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective single-arm study with historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Robotic CME (Experimental): Robot-assisted extended right colectomy
  Interventions: Device: Robot-assisted laparoscopic extended right colectomy

INTERVENTIONS:
Device: Robot-assisted laparoscopic extended right colectomy — An extended right hemicolectomy with total mesocolic excision and meticulous central dissection as described by Hohenberger will be performed with the DaVinci Xi robot by one of two dedicated surgeons
  Other Names: DaVinci Xi

SUMMARY:
A single-center prospective study to elucidate whether extended robot-assisted right colectomy (e-RARC) performs as well as extended open right colectomy (e-ORC) in terms of specimen quality, and in addition, whether less postoperative morbidity and shorter length of stay (LOS) can be attained. Patients with colonic cancer near the right flexure or the oral part of the transverse colon will be compared excluding the most technically demanding and frail patients in both groups. A total of 40 patients undergoing e-RARC in a prospective series will be included and compared with 44 consecutive patients previously treated with e-ORC.

DETAILED DESCRIPTION:
Complete mesocolic excision with central vascular ligation (CME) is an improvement of surgical technique in the operation for colonic cancer suggested to increase long-term survival. The concept was originally developed for open surgery by W. Hohenberger in Erlangen with excellent survival rates. However, if the tumor is located in the transverse colon or near the right colonic flexure, the procedure is particularly technically demanding, and for that reason most surgeons still prefer to do it by open operation (laparotomy) instead of the minimally invasive approach (laparoscopy) presently recommended for colonic cancer surgery. The advent of robotic surgery has improved the dexterity of instruments used in laparoscopic surgery and pushed the limits of what is possible with a minimally invasive approach. Since minimally invasive surgery is associated with better outcomes in terms of postoperative morbidity, pain, length of stay etc., it would be highly desirable if CME surgery could be done by robot-assisted laparoscopic operation instead of the current open approach. The current single-center study is proposed to elucidate whether extended robot-assisted right colectomy (e-RARC) performs as well as extended open right colectomy (e-ORC) in terms of specimen quality, and in addition, whether less postoperative morbidity and shorter length of stay (LOS) can be attained. Patients with colonic cancer near the right flexure or the oral part of the transverse colon will be compared excluding the most technically demanding and frail patients in both groups. A total of 40 patients undergoing e-RARC in a prospective series will be included and compared with 44 consecutive patients previously treated with e-ORC.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or verified colonic cancer visualized by colonoscopy and on CT in the anal part of the ascending colon, in the right flexure or in the oral 2/3 of the transverse colon
* Patient is 18 years or older, legally competent and able to comprehend information and give consent
* Tumor is UICC stage I-III on preop CT
* Operation is elective

Exclusion Criteria:

* Previous major open intraabdominal surgery
* Ileus or other acute abdominal condition
* CT scan with suspicion of T4 tumor
* RITA score > 3 (Preop risk and frailty score)
* BMI > 35 kg/m2
* Project surgeon not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Plane of dissection | 30 days
  As judged by pathologist (mesocolic/intramesocolic/intramuscular)
Lymph node count | 30 days
  Number of nodes in specimen, as determined by pathologist

SECONDARY OUTCOMES:
Complications | 30 days
  Postoperative complications, graded by Clavien-Dindo
Reinterventions | 30 days
  Reinterventions under anesthesia before discharge from hospital
Length of stay | 30 days
  Days from operation to discharge from hospital
Readmissions | 30 days
  Readmissions to hospital 1-30 days after initial discharge

OTHER OUTCOMES:
Operation time | intraoperative
  Minutes from first incision to final stitch
Conversion rate | 30 days
  Percentage of conversions from robotic to open surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bundgaard, MD, Principal Investigator — Department of Surgery
Locations (1):
- Vejle Hospital, Department of Surgery, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No